CLINICAL TRIAL: NCT05280132
Title: Use of MULTIplex PCR, Procalcitonin, and Sputum Appearance to Reduce Duration of Antibiotic Therapy During Severe COPD EXAcerbation: A Controlled, Randomized, Open-label, Parallel-Group, Multicenter Trial
Acronym: MULTI-EXA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP210085; 2021-005435-23 (EudraCT Number)
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-03

CONDITIONS: Acute Exacerbation of COPD
Keywords: AECOPD; respiratory multiplex PCR; Appearance of sputum; Procalcitonin; Antibiotics saving; Diagnosis; Treatment
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized strategy (Experimental): Personalized antibiotic treatment based on mPCR results, PCT (values and kinetics) and appearance of sputum.
  A broad panel respiratory mPCR FA-PPP is performed on a respiratory tract sample collected 12 hours after inclusion.
  After inclusion (D0), an algorithm of early antibiotic adaptation and discontinuation will be applied immediately and repeated every day until day 7.
  This algorithm of early antibiotic adaptation and discontinuation is based on a multimodal approach, using:
  * The appearance of sputum (clinical approach);
  * PCT values and kinetics (biological approach);
  * Results of mPCR FA-PPP (microbiological approach).
  Interventions: Procedure: Personalized antibiotic treatment
- Usual strategy (Other): Usual antibiotic treatment
  Left at the discretion of the physician as in usual practice
  Interventions: Other: Usual antibiotic treatment

INTERVENTIONS:
Procedure: Personalized antibiotic treatment — Personalized antibiotic treatment based on mPCR results, PCT (values and kinetics) and appearance of sputum.
  Arms: Personalized strategy
Other: Usual antibiotic treatment — The antimicrobial therapy is left at the discretion of the physicians, as in usual practice.
  Arms: Usual strategy

SUMMARY:
COPD is a common chronic disease. Its natural course is characterized by Acute exacerbations (AE). This may require hospitalization or even ICU/RESUSCITATION admission. The most common causes are respiratory distress with hypercapnic acidosis that requires mechanical ventilation (Invasive or non-invasive). Lower respiratory tract infections, bacteria and/or viruses are the main pathogenic factors of AE. The treatment of AECOPD is initially symptomatic treatment, combining bronchodilators, ventilatory support (oxygen therapy and/or mechanical ventilation) and respiratory physiotherapy. Systemic corticosteroid therapy is optional. When i) the sputum is purulent and ii) increased dyspnea and / or an increase in sputum volume is observed, antibiotic treatment is recommended for hospitalized patients. Antibiotic therapy is routinely recommended when mechanical ventilation is required.

During ICU/RESUSCITATION AECOPD, more than 85% of patients received antibiotic therapy, with a median duration of 8 to 9 days, and the benefit of antibiotic therapy is likely to be limited to infected patients. Suspected or documented lower respiratory tract bacteria, that is, 25% to 50% of patients. This will lead to overuse of antibiotics, which is a problem for patients and the community.

A personalized antibiotic strategy could limit this phenomenon, relying on multimodal methods, using aspect of sputum (clinical method), procalcitonin (PCT) (biological method) and the FilmArray ™ Pneumonia Panel extended panel multiplex respiratory PCR Plus (mPCR FA-PPP) (Biomérieux®) (microbiological approach).

The hypothesis of this study is that sputum appearance, procalcitonin (PCT) and the FilmArray ™ Pneumonia Panel Plus expanded panel multiplex respiratory PCR (mPCR FA-PPP) (Biomérieux®) could be used in combination , and their results integrated into a decision-making algorithm aimed at personalizing antibiotic therapy and guiding its early termination in patients admitted to ICU/RESUSCITATION due to acute exacerbation of chronic obstructive pulmonary disease (AECOPD) to the main benefit of antibiotic savings, and without additional risk to patient safety.

DETAILED DESCRIPTION:
Inclusion (D0_H0) is performed in ICU/RESUSCITATION. The interval between admission to the hospital and admission to ICU/RESUSCITATION must be maximum 72 hours. Conventional microbiological investigations are left at the discretion of the physicians, and may include blood cultures, L. pneumophila and S. pneumoniae antigens. Usual biology includes procalcitonin measurement. Empirical antimicrobial therapy must be started as soon as possible after inclusion.

Randomization is performed immediately after the inclusion. In the intervention arm, a broad panel respiratory mPCR FA-PPP is performed on respiratory tract sample (tracheal aspirate, BAL or sputum), collected 12 hours after inclusion. An algorithm of early antibiotic adaptation and discontinuation, based on the microbiological results, including the mPCR FA-PPP results, and the procalcitonin values and kinetics and also aspect of sputum will be used. This algorithm will be applied as soon as possible after inclusion, and repeated day after day until D7.

In the control arm, the antimicrobial therapy is left at the discretion of the physicians, as in usual practice.

Evaluation criteria are collected at hospital discharge or at D28, and D90. The vital status may be obtained by phone call at D28 (if the patient has been discharged before D28) and at D90.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* COPD (according to GOLD 2020), whatever the stage (I-IV)
* Acute exacerbation (defined as the onset or worsening of one or more of the usual signs/symptoms of COPD) with acute worsening of respiratory symptoms that result in additional therapy) with acute respiratory failure requiring admission to ICU and ventilatory support (invasive mechanical ventilation or non-invasive mechanical ventilation or high-flow nasal oxygen therapy with FiO2 ≥ 50%)
* Informed consent of patient, patient's immediate family/ or inclusion in an emergency situation
* Affiliation to a social security

Exclusion Criteria:

* The interval between admission to the hospital and admission to ICU more than 3 days
* Antibiotic therapy clearly needed for a suspected or documented extra-respiratory infection
* Congenital or acquired immunosuppression (congenital immune deficiency, high-grade hematologic malignancies, use of immunosuppressive drugs in the last 30 days including anti-cancer chemotherapy and antirejection medications, corticosteroid treatment ≥ 20 mg/d prednisone equivalent for at least 14 days, neutropenia, HIV with unknown or known CD4 <200 / µL in the past 6 months)
* Tracheotomy
* Bronchiectasis / cystic fibrosis
* Moribund patient (imminent death)
* Patient deprived of liberty and / or under legal protection measure
* Patient already included in MULTI-EXA
* Patient already included in a type 1 interventional study on antibiotics
* Ongoing pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of antibiotic-free days | Day 28
  The number of days alive without antibiotics at Day 28.

SECONDARY OUTCOMES:
Number of days with antibiotics in survivors at D28 | Day 28
Number of days with broad spectrum antibiotics in survivors at D28 | Day 28
Nosocomial pneumonia incidence rate | Day 28
Multidrug-resistant bacteria colonization / infection rate | Day 28
ICU lengths of stay | Day 28
Hospital lengths of stay | Day 28
Number of days alive without mechanical ventilation (invasive or non-invasive) | Day 28
Incidence rates of Hospital-acquired pneumonia (including ventilator-associated pneumonia) | Day 28
Mortality rates (in ICU, in hospital) | Day 28 and Day 90
Number of additional AECOPD (requiring hospitalization and / or initiation of systemic corticosteroid therapy and / or antibiotic therapy) after the initial AECOPD | Day 90
Time between the initial AECOPD and the following AECOPD (AECOPD requiring hospitalization and / or initiation of systemic corticosteroid therapy and / or antibiotic therapy) | Day 90
COPD-related symptoms | Day 90
  Using the COPD Assessment Test (CAT) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume VOIRIOT, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Intensive care department-Hospital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-participant data will be made available outside the primary research group for secondary research purposes like re-analysis, secondary analysis, or meta-analysis, and shared via an online secured platform.